CLINICAL TRIAL: NCT02401867
Title: Preventive Sexual Health Screening Among Female-to-Male (FTM) Transgender Adult Patients
Status: Completed | Type: Observational
Sponsor: Fenway Community Health (Other)
Collaborators: Patient-Centered Outcomes Research Institute (Other)
Responsible Party: Principal Investigator, Sari Reisner, ScD, Research Scientist, Fenway Community Health
Other Study IDs: CER-1403-12625
Record Dates: First submitted 2015-01-30; First posted 2015-03-30 (Estimated); Results first posted 2017-06-28 (Actual); Last update posted 2017-06-28 (Actual); Status verified 2017-04

CONDITIONS: Uterine Cervical Neoplasms; Sexually Transmitted Diseases
Keywords: transgender; female-to-male; cervical cancer; HPV; sexual health
MeSH Terms: conditions — Uterine Cervical Neoplasms; Sexually Transmitted Diseases

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to assess the acceptability and effectiveness of utilizing vaginal self-swabs for HPV DNA testing as compared to provider-collected cervical swabs for HPV, as well as to investigate the prevalence of other Sexually Transmitted Infections (STIs) among sexually active female-to-male (FTM) transgender adults.

DETAILED DESCRIPTION:
This observational study will examine sexual health in a bio-behavioral cross-sectional mixed-methods design among 150 FTM patients in Boston, Massachusetts, and will determine the acceptability as well as collect epidemiologic data on the comparative performance characteristics of several biological screening modalities in this patient population. Patients and stakeholders are key partners throughout the project and are involved in all phases of study development, implementation, and plans for dissemination.

Eligible participants will participate in a one-time clinical visit. Following written consent, the one-time clinical visit will include: 1) Quantitative assessment; 2) Collection of biological specimens/biomarkers (HPV DNA vaginal self-swab, HPV DNA cervical swab collected by provider, Pap test with cytology, STI testing self- and provider-collected); 3) Qualitative Interview.

A series of national, online focus groups with FTMs, providers, and key stakeholders will occur to gather information on the sexual health needs of FTM individuals outside the Boston area and to ensure that the dissemination of study findings take differing demographic concerns into consideration.

ELIGIBILITY:
Inclusion Criteria:

* Age 21-64
* Assigned a female sex at birth and now self-identifies as a man, trans masculine, trans man, FTM, transgender, genderqueer/non-binary, transsexual, male, and/or another diverse transgender identity or expression
* Have a cervix
* Sexually active in the past 36 months (with sexual partner(s) of any gender)
* Able to speak and understand English
* Willing and able to provide informed consent

Exclusion Criteria:

* Unable to provide informed consent due to severe mental or physical illness
* Substance intoxication at the time of interview

Ages: 21 Years to 64 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: This study aims to enroll 150 female-to-male (FTM) individuals, ages 21-64. Participants will be recruited from the existing FTM patient population at Fenway Health, as well as via community outreach in the greater Boston area. A diverse sample is anticipated; the aim is to recruit 40% racial/ethnic minority FTMs.
Sampling Method: Probability Sample
Enrollment: 150 (Actual)
Dates: Start 2015-01; Primary Completion 2016-09 (Actual); Study Completion 2016-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sari Reisner, ScD, Principal Investigator — Fenway Community Health
Locations (1):
- Fenway Community Health, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Suarez NA, Peitzmeier SM, Potter J, Samandur A, Reisner SL. Preliminary findings for adverse childhood experiences and associations with negative physical and mental health and victimization in transmasculine adults. Child Abuse Negl. 2021 Aug;118:105161. doi: 10.1016/j.chiabu.2021.105161. Epub 2021 Jun 16. PMID 34146966
- [Derived] Pletta DR, White Hughto JM, Peitzmeier S, Deutsch MB, Pardee D, Potter J, Reisner SL. Individual- and Partnership-Level Correlates of Protective Barrier Use in a Sample of Transmasculine Adults with Diverse Sexual Partnerships. AIDS Patient Care STDS. 2020 May;34(5):237-246. doi: 10.1089/apc.2019.0296. PMID 32396475
- [Derived] McDowell MJ, Hughto JMW, Reisner SL. Risk and protective factors for mental health morbidity in a community sample of female-to-male trans-masculine adults. BMC Psychiatry. 2019 Jan 9;19(1):16. doi: 10.1186/s12888-018-2008-0. PMID 30626372
- [Derived] Agenor M, White Hughto JM, Peitzmeier SM, Potter J, Deutsch MB, Pardee DJ, Reisner SL. Gender identity disparities in Pap test use in a sample of binary and non-binary transmasculine adults. J Gen Intern Med. 2018 Jul;33(7):1015-1017. doi: 10.1007/s11606-018-4400-3. No abstract available. PMID 29654599
- [Derived] Reisner SL, Deutsch MB, Peitzmeier SM, White Hughto JM, Cavanaugh T, Pardee DJ, McLean S, Marrow EJ, Mimiaga MJ, Panther L, Gelman M, Green J, Potter J. Comparing self- and provider-collected swabbing for HPV DNA testing in female-to-male transgender adult patients: a mixed-methods biobehavioral study protocol. BMC Infect Dis. 2017 Jun 23;17(1):444. doi: 10.1186/s12879-017-2539-x. PMID 28645254

RESULTS

PARTICIPANT FLOW:
Groups:
- Overall Sample: Overall sample reported as all participants received both the self and the provider swab.
Period: Enrolled
Arm/Group | Overall Sample
Started | 150
Completed | 150
Not Completed | 0
Period: Specimen Collection
Arm/Group | Overall Sample
Started | 150
Completed | 140 (Completed both vaginal self-swab and provider-collected cervical swab)
Not Completed | 10
Not completed — Didn't receive 1 or more tests | 10
Period: Analysis
Arm/Group | Overall Sample
Started | 140
Completed | 131 (Comparative analysis of vaginal HPV DNA results and cervical HPV DNA results)
Not Completed | 9
Not completed — Cervical assay could not be conducted | 9

BASELINE CHARACTERISTICS:
Population: Enrolled =150, analytic sample =131: 10 participants did not receive the vaginal HPV DNA self-swab and provider cervical swab; 7 received the self-swab, but not the provider; 1 received the provider-swab, but not the self; and 2 did not receive either test. Additionally, 9 of the provider samples could not be assayed due to low cellular content.
Groups:
- Full Sample: Descriptive characteristics for the full sample (n=150).
Arm/Group | Full Sample
Number analyzed (Participants) | 150
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 150
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 27.49 (5.74)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Trans Masculine/ Male to Female | 150
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 9
  Native Hawaiian or Other Pacific Islander | 1
  Black or African American | 4
  White | 112
  More than one race | 23
  Unknown or Not Reported | 1
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Yes, Hispanic/Latino | 14
  Not Hispanic/Latino | 133
  Unknown | 3
Region of Enrollment [Number; unit: participants]
  United States | 150
Diagnosed with Chlamydia - Lifetime [Count of Participants; unit: Participants]
  Yes | 8
  No | 142
Diagnosed with Gonorrhea - Lifetime [Count of Participants; unit: Participants]
  Yes | 5
  No | 145
Diagnosed with Syphilis - Lifetime [Count of Participants; unit: Participants]
  Yes | 1
  No | 149
Diagnosed with Trichomoniasis - Lifetime [Count of Participants; unit: Participants]
  Yes | 6
  No | 144
Diagnosed with Hepatitis C - Lifetime [Count of Participants; unit: Participants]
  Yes | 1
  No | 149
Diagnosed with Genital Herpes - Lifetime [Count of Participants; unit: Participants]
  Yes | 5
  No | 145
Diagnosed with Genital Warts - Lifetime [Count of Participants; unit: Participants]
  Yes | 4
  No | 146
Diagnosed with HPV - Lifetime [Count of Participants; unit: Participants]
  Yes | 11
  No | 135
  Don't Know | 3
  Prefer Not to Answer | 1
HIV Status - Lifetime [Count of Participants; unit: Participants]
  Positive | 1
  Negative | 120
  Don't Know | 28
  Prefer Not to Answer | 1
Provider-Collected Cervical Cytology (Current) [Count of Participants; unit: Participants]
  Abnormal | 9
  Normal | 111
  Assay could not be tested | 27
  Assay not collected | 3
Provider-Collected Cervical HPV DNA (Current) [Count of Participants; unit: Participants]
  Positive | 21
  Negative | 111
  Assay could not be tested | 9
  Assay not collected | 9
Self-Collected Vaginal HPV DNA (Current) [Count of Participants; unit: Participants]
  Positive | 21
  Negative | 126
  Assay not collected | 3

OUTCOME MEASURES:

1. Primary Outcome: Concordance Between Vaginal Self-swab Results and Provider-collected Cervical Swab Results for HPV DNA Among Sexually Active FTM Adults
Description: Quantitatively assessed the non-inferiority of vaginal self-swab for HPV DNA compared to provider-collected cervical swab for HPV via laboratory confirmed testing in sexually active FTM adults. Compared the concordance of the positive self-swab HPV DNA test results to the positive cervical provider swab HPV DNA test results (reference) using the McNemar's test, a two-sample test for binomial proportions for matched-pair data.
Time Frame: 1 day
Population: Analytic sample =131: 10 participants did not receive both the vaginal self-swab HPV DNA test and the provider cervical test (reference); 7 received the self, but not the provider; 1 received the provider, but not the self; 2 did not receive either test. Additionally, 9 of the provider samples could not be assayed due to low cellular content.
Measure: Count of Participants; unit: Participants
Groups:
- Participants With Positive Cervical HPV DNA Test Result: Positive result determined by reference test: provider cervical HPV DNA Hybridization assay
- Participants With a Negative Cervical HPV DNA Test Result: Negative result determined by reference test: provider cervical HPV DNA Hybridization assay
Arm/Group | Participants With Positive Cervical HPV DNA Test Result | Participants With a Negative Cervical HPV DNA Test Result
Number analyzed (Participants) | 21 | 110
Participants
  Positive vaginal self-swab HPV DNA test | 15 | 2
  Negative vaginal self-swab HPV DNA test | 6 | 108
Statistical Analysis 1: Comparison: Participants With Positive Cervical HPV DNA Test Result vs Participants With a Negative Cervical HPV DNA Test Result; Comparing the concordance of the HPV DNA-positive results to the cervical provider swab HPV DNA test results (reference) using the McNemar's test, a two-sample test for binomial proportions for matched-pair data. Null hypothesis: The sensitivities between swab 1 (self-vaginal) and swab 2 (provider-cervical) are equal [ H0 : p1 = p2 ]; Test type: Non-Inferiority or Equivalence — We selected our initial sample size of 150 participants to detect a clinically meaningful % discordance between the two sampling approaches and achieve 90% power at the 0.05 alpha-level using McNemar's test adjusted for analysis of clustered matched-pair data; p = .29, McNemar — Statistical significance was determined at an a priori threshold of p <0.05; Degrees of freedom = 1
Statistical Analysis 2: Comparison: Participants With Positive Cervical HPV DNA Test Result vs Participants With a Negative Cervical HPV DNA Test Result; Concordance of HPV DNA detection between self-swab and provider swab assessed via an unweighted Kappa (K) statistic to determine the percentage agreement beyond that expected by chance; Test type: Superiority or Other; p < 0.001, Kappa — A priori threshold: p<0.05; Kappa = .75, 95% CI 2-sided [0.58 to 0.92], Standard Error of Mean 0.08 — Using the asymptotic standard error assuming the null hypothesis
Statistical Analysis 3: Comparison: Participants With Positive Cervical HPV DNA Test Result; Assessed sensitivity of vaginal self-swab HPV DNA with respect to provider cervical HPV DNA (reference test); Test type: Superiority or Other; Sensitivity = 71.43, 95% CI 2-sided [47.82 to 88.72] — Used exact confidence intervals
Statistical Analysis 4: Comparison: Participants With a Negative Cervical HPV DNA Test Result; Test type: Non-Inferiority or Equivalence — Assessed specificity of vaginal self-swab HPV DNA with respect to provider cervical HPV DNA (reference test); Specificity = 98.18, 95% CI 2-sided [93.59 to 99.78] — Used exact confidence intervals
Statistical Analysis 5: Comparison: Participants With Positive Cervical HPV DNA Test Result; Assessed positive predictive value of vaginal self-swab HPV DNA with respect to provider cervical HPV DNA (reference test); Test type: Superiority or Other; Positive Predictive Value = 88.24, 95% CI 2-sided [63.56 to 98.54] — Used exact confidence intervals
Statistical Analysis 6: Comparison: Participants With a Negative Cervical HPV DNA Test Result; Assessed negative predictive value of vaginal self-swab HPV DNA with respect to provider cervical HPV DNA (reference test); Test type: Superiority or Other; Negative predictive value = 94.74, 95% CI 2-sided [88.90 to 98.04] — Used exact confidence intervals

ADVERSE EVENTS:
Arm/Group | Full Sample
Serious Adverse Events (participants affected / at risk) | 0/150
Other Adverse Events (participants affected / at risk) | 0/150

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days